CLINICAL TRIAL: NCT04936061
Title: A Transnasal Evaporative Cooling Device for Acute Treatment of Migraine
Brief Title: Transnasal Cooling for Migraine
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment problems
Sponsor: CoolTech LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P-224011-0040
Record Dates: First submitted 2021-06-15; First posted 2021-06-23 (Actual); Results first posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Migraine; Episodic Migraine; Migraine With Aura; Migraine Without Aura
MeSH Terms: conditions — Migraine Disorders; Migraine with Aura; Migraine without Aura

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- High flow treatment (Experimental): 15 minute transnasal air flow therapy with the CoolStat active device as an abortive treatment for migraine attack.
  Interventions: Device: CoolStat active device
- Low flow treatment (Experimental): 15 minute transnasal air flow therapy with the CoolStat active device as an abortive treatment for migraine attack.
  Interventions: Device: CoolStat active device
- Sham flow ambient air (Sham Comparator): 15 minute transnasal air flow therapy with the CoolStat sham device as an abortive treatment for migraine attack.
  Interventions: Device: CoolStat sham device

INTERVENTIONS:
Device: CoolStat active device — The CoolStat active device will administer a therapeutic flow of dry air into the nostril.
  Arms: High flow treatment; Low flow treatment
Device: CoolStat sham device — The CoolStat sham device will administer a sham flow of ambient air into the nostril.
  Arms: Sham flow ambient air

SUMMARY:
This is a prospective, double-blind, sham-controlled, randomized study to assess the safety, tolerability, and optimal dose of the COOLSTAT Transnasal Thermal Regulating Device for acute treatment of migraine. The hypothesis is that evaporative cooling induced by the CoolStat using only ambient, dry air will reduce the pain and other symptoms of migraine headaches during an acute migraine episode.

ELIGIBILITY:
Inclusion Criteria:

1. Meets the International Classification of Headache Disorders (ICHD-3) diagnostic criteria for migraine with or without aura, with the exception of ''complicated migraine'' (i.e., hemiplegic migraine, ophthalmoplegic migraine, migrainous infarction).
2. Patient is between 18 and 80 years of age.
3. Patient experiences 2 to 8 migraine attacks per month.
4. Patient is in good reported general health, with no fever (<38.3C/101F).
5. Patient has had diagnosis of migraine with or without aura over at least 1 year.
6. Migraine onset before 50 years of age.
7. Migraine prophylaxis medication unchanged for 6 weeks prior to study enrollment.
8. Able to attend treatment session within 6 hours of migraine onset, with 48 hours of pain freedom prior to onset of migraine attack.
9. Migraine pain severity of Grade 2 or Grade 3 on day of treatment.
10. Provision of signed and dated informed consent form.
11. Stated willingness to comply with all study procedures and availability for the duration of the study.

Exclusion Criteria:

1. has difficulty distinguishing his or her migraine attacks from tension-type headaches
2. Patient has uncontrolled hypertension.
3. Patient has a fever (≥38.3C / 101F).
4. Patient has used opioid medication or barbiturates in the past month.
5. Patient has Medication Overuse Headache (MOH), New Daily Persistent Headache (NDPH) or Chronic Tension Type Headache (CTTH).
6. Patient has 15 or more headache days per month.
7. Patient has used acute treatment(s) for migraine in the 48 hours preceding treatment i.e. over-the-counter (OTC) medications, prescription medications, or medical device).
8. Patient has received Botox treatment, supraorbital or occipital nerve blocks in the last 4 weeks.
9. Intolerance to intranasal neurostimulation or sensory processing disorder that makes the treatment not applicable.
10. Recurrent epistaxis or chronic rhinosinusitis.
11. Recent facial trauma, sinus or intranasal surgery within the last 4 months.
12. Known or suspected pregnancy.
13. Unable to fully understand the consent process and provide informed consent due to either language barriers or mental capacity.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nauman Tariq, MD, Principal Investigator — Atrium Health Neurosciences Institute
Locations (3):
- United States (3):
  - Mayo Clinic, Scottsdale, Arizona
  - Michigan State University, East Lansing, Michigan
  - Atrium Health Neurosciences Institute, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 87 subjects consented, 24 of whom were randomized to a treatment group. 63 subjects did not return to study sites for randomization during an active migraine attack during the 60-day enrollment period. 7 of those subjects reconsented for an additional 60- day enrollment period. Only two subjects who reconsented came to the clinic for randomization. 4 subjects were withdrawn post-consent because they became in eligible (3) or withdrew their consent (1).
Period: Overall Study
Arm/Group | High Flow Treatment | Low Flow Treatment | Sham Flow Ambient Air
Started | 6 | 9 | 9
Completed | 6 | 9 | 9
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Flow Treatment | Low Flow Treatment | Sham Flow Ambient Air | Total
Number analyzed (Participants) | 6 | 9 | 9 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 8 | 8 | 22
  >=65 years | 0 | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] — Subjects provided their age at time of enrollment on screening questionnaire.
  years | 37.8 (12.3) | 51.4 (13.2) | 50.3 (9.7) | 47.6 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 9 | 24
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 9 | 8 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 3
  White | 5 | 8 | 7 | 20
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 9 | 9 | 24

OUTCOME MEASURES:

1. Primary Outcome: Pain Relief
Description: The percentage of patients having a reduction of a moderate or severe migraine headache (Grade 2 or 3) at baseline to a mild headache or to no headache (Grade 1 or 0) at 2 hours after the CoolStat treatment session.
Time Frame: 2 hours
Population: The primary analysis was based on a mixed logistic regression model using the variable Pain Relief without rescue medication at 2 hours post treatment as the outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | High Flow Treatment | Low Flow Treatment | Sham Flow Ambient Air
Number analyzed (Participants) | 6 | 9 | 9
Participants | 3 | 4 | 8

2. Primary Outcome: Tolerability of the CoolStat Device
Description: Number of subjects who fail to complete the full treatment session
Time Frame: 15 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | High Flow Treatment | Low Flow Treatment | Sham Flow Ambient Air
Number analyzed (Participants) | 6 | 9 | 9
Participants | 2 | 1 | 0

3. Primary Outcome: Safety of the CoolStat Device
Description: Number of participants with device-related adverse events
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | High Flow Treatment | Low Flow Treatment | Sham Flow Ambient Air
Number analyzed (Participants) | 6 | 9 | 9
Participants | 3 | 3 | 0

4. Secondary Outcome: Pain Relief
Description: The percentage of patients having a reduction of a moderate or severe migraine headache (Grade 2 or 3) at baseline to a mild headache or to no headache (Grade 1 or 0) immediately after the CoolStat treatment session.
Time Frame: 0 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | High Flow Treatment | Low Flow Treatment | Sham Flow Ambient Air
Number analyzed (Participants) | 6 | 9 | 9
Participants | 0 | 3 | 7

5. Secondary Outcome: Pain Relief
Description: The percentage of patients having a reduction of a moderate or severe migraine headache (Grade 2 or 3) at baseline to a mild headache or to no headache (Grade 1 or 0) at 24 hours after the CoolStat treatment session without the use of rescue medication
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | High Flow Treatment | Low Flow Treatment | Sham Flow Ambient Air
Number analyzed (Participants) | 6 | 9 | 9
Participants | 1 | 2 | 5

6. Secondary Outcome: Pain Freedom
Description: The percentage of patients having a reduction of a moderate or severe migraine headache (Grade 2 or 3) at baseline to no headache (Grade 0) at 2 hours after the CoolStat treatment session without the use of rescue medication
Time Frame: 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | High Flow Treatment | Low Flow Treatment | Sham Flow Ambient Air
Number analyzed (Participants) | 6 | 9 | 9
Participants | 0 | 0 | 4

7. Secondary Outcome: Pain Freedom
Description: The percentage of patients having a reduction of a moderate or severe migraine headache (Grade 2 or 3) at baseline to no headache (Grade 0) at 24 hours after the CoolStat treatment session without the use of rescue medication.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | High Flow Treatment | Low Flow Treatment | Sham Flow Ambient Air
Number analyzed (Participants) | 6 | 9 | 9
Participants | 1 | 0 | 4

8. Secondary Outcome: Relief From Migraine-associated Symptoms
Description: The percentage of patients having a reduction in symptom severity from Grade 3/2 at baseline to Grade 1/0 at 2 hours post-treatment session without the use of rescue medication.
Time Frame: 2 hours
Population: Most Bothersome Symptom scores at baseline and at 2 hours post treatment were compared for this analysis
Measure: Count of Participants; unit: Participants
Arm/Group | High Flow Treatment | Low Flow Treatment | Sham Flow Ambient Air
Number analyzed (Participants) | 6 | 9 | 9
Participants | 4 | 6 | 7

9. Secondary Outcome: Freedom From Migraine-associated Symptoms
Description: The percentage of patients with absence of photophobia, phonophobia, nausea and vomiting, at 2 hours after the end of the CoolStat treatment session without the use of rescue medication
Time Frame: 2 hours
Population: Most Bothersome Symptom scores at baseline and at 2 hours post treatment were compared for this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | High Flow Treatment | Low Flow Treatment | Sham Flow Ambient Air
Number analyzed (Participants) | 6 | 9 | 9
Participants | 3 | 3 | 5

10. Secondary Outcome: Use of Rescue Medication
Description: The percentage of patients who took acute anti-migraine medication within 24 hours after the end of the CoolStat treatment session.
Time Frame: 0 to 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | High Flow Treatment | Low Flow Treatment | Sham Flow Ambient Air
Number analyzed (Participants) | 6 | 9 | 9
Participants | 4 | 8 | 4

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | High Flow Treatment | Low Flow Treatment | Sham Flow Ambient Air
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 3/6 | 3/9 | 0/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Flow Treatment (N=6) | Low Flow Treatment (N=9) | Sham Flow Ambient Air (N=9)
Burning sensation in nostril (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Increased head pain (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (General disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-02): https://cdn.clinicaltrials.gov/large-docs/61/NCT04936061/Prot_SAP_000.pdf